CLINICAL TRIAL: NCT01581242
Title: A Randomized, Open-label, Three-sequence, Three-period, Three-treatment Clinical Trial to Investigate the Pharmacokinetic Drug-drug Interaction of Clevudine and Adefovir Dipivoxil After Oral Administration in Healthy Male Subjects
Brief Title: A Clinical Trial to Investigate the Pharmacokinetic Drug-drug Interaction of Clevudine and Adefovir Dipivoxil After Oral Administration in Healthy Male Subjects
Acronym: BKP-1003-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKP-1003
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Clevudine and Adefovir dipivoxil; pharmacokinetic drug drug interaction; oral administration; male subjects
MeSH Terms: interventions — clevudine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Clevudine, Adefovir dipivoxil , Clevudine+Adefovir dipivoxil
- B (Experimental)
  Interventions: Drug: Clevudine; Adefovir dipivoxil ,Clevudine +Adefovir dipivoxil
- C (Experimental)
  Interventions: Drug: Clevudine,Adefovir dipivoxil ,Clevudine +Adefovir dipivoxil

INTERVENTIONS:
Drug: Clevudine, Adefovir dipivoxil , Clevudine+Adefovir dipivoxil — Clevudine 20mg qd Days 1; Adefovir dipivoxil 10 mg qd Days 8;Clevudine 20mg +Adefovir dipivoxil 10mg qd Days 15
  Arms: A
Drug: Clevudine; Adefovir dipivoxil ,Clevudine +Adefovir dipivoxil — Clevudine 20mg +Adefovir dipivoxil 10mg qd Days 1; Clevudine 20mg qd Days 8; Adefovir dipivoxil 10 mg qd Days 15;
  Arms: B
Drug: Clevudine,Adefovir dipivoxil ,Clevudine +Adefovir dipivoxil — Adefovir dipivoxil 10 mg qd Days 1;Clevudine 20mg +Adefovir dipivoxil 10mg qd Days 8; Clevudine 20mg qd Days 15
  Arms: C

SUMMARY:
This is a randomized, open-label, three-sequence, three-period, three-treatment clinical trial to investigate the pharmacokinetic drug-drug interaction of Clevudin and Adefovir dipivoxil after oral administration in healthy male subjects.

DETAILED DESCRIPTION:
To evaluate the safety, drug-tolerance, pharmacokinetics of Clevudine or Adefovir monotherapy or Adefovir and Clevudine combination in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Age limit is from 20 to 45 with healthy male subjects in screening
* Weight limit is from 50kg(110.23Ib) to 90kg(198.41Ib) with BMI 18.5-26 (BMI(kg/m2)= weight(kg)/{height(m)}2
* The person who fully understands and listens about this clinical trial, receives written consent to observe the notandum and decides to participate voluntarily

Exclusion Criteria:

* The person who has past history or serious disease in liver, kidney, nervous system, respiratory system, gastro-intestinal tract system, endocrine system, blood tumor, cardio-vascular system, urinary system, mental system clinically
* The person who has the past history of Gastro-intestinal operation(except simple appendectomy or herniotomy)or Gastro-intestinal system disease (Chron's disease,ulcer,acute and chronic pancreatitis, etc) that can be influenced the absorption of clinical drug
* The person who has the past history of hypersensitivity reaction about the drugs that contain the identical affiliation ingredient or ingredient of Clevudine, Adefovir dipivoxil or others drugs(aspirin, antibiotics etc)or has the significant past history of hypersensitivity reaction clinically
* The person who shows results of the 1.5 times upper limit in screening test of AST(SGOT), ALT(SGPT)
* The person who shows results of the positive HBsAg, HCV Ab,HIV Ab
* The person who has a past history of drug abuse or shows a positive result of drug abuse in urine drug analysis of screening test
* The person who takes medications of some medicine and medical supplies or oriental medicine within 2 weeks before the first administration date', or some OTC drug, vitamin supplements or health functional food within 1week (if only,it's confirmed by the investigator's judgment that they are not affected in pharmacokinetics character and safety evaluation about the clinical drugs)
* The person who participates in other clinical trials within 2 weeks before the first administration date'
* The person who donates plasma pheresis within 1 month before the first administration date, donates whole blood within 2 months before the first administration date or receives a transfusion within a month before the first administration date
* Persistent drinker(over 21 units/week, 1 unit = 10g of pure alcohol) or a drinker who can't stop drinking during hospitalization period
* Smoker who takes a drag over 10 cigarettes per day during the past three months
* The person who was judged unfit for participating in clinical trials by a investigator because of the clinical laboratory test results or other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
AUClast | Predose ~24hrs
Cmax | Predose~24hrs

SECONDARY OUTCOMES:
AUCinf | Predose~24hrs
Tmax | Predose~24hrs
T1/2 | Predose~24hrs
CL/F | Predose~24hrs
Safety | Screening, predose, post 24h, Post-study visit
  clinically measured adverse events, abnormality of laboratory tests abnormality of vital signs,ECG e.t.c

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea